CLINICAL TRIAL: NCT01905215
Title: An Observer-blind Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Respiratory Syncytial Virus (RSV) Investigational Vaccine (GSK3003891A) in Healthy Men
Brief Title: Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Investigational Respiratory Syncytial Virus (RSV) Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 116969
Record Dates: First submitted 2013-07-11; First posted 2013-07-23 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infections, Respiratory Syncytial Virus
Keywords: Immunogenicity; Respiratory Syncytial Virus; Reactogenicity; Vaccination; Safety
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (8):
- Group A (Experimental): Subjects in this group will receive a single dose of formulation 1 of RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003892A (formulation 1)
- Group B (Experimental): Subjects in this group will receive a single dose of formulation 2 of RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003893A (formulation 2)
- Group C (Experimental): Subjects in this group will receive a single dose of formulation 3 of RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003895A (formulation 3)
- Group D (Experimental): Subjects in this group will receive a single dose of formulation 4 of RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003896A (formulation 4)
- Group E (Experimental): Subjects in this group will receive a single dose of formulation 5 of RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003898A (formulation 5)
- Group F (Experimental): Subjects in this group will receive a single dose of formulation 6 of RSV vaccine
  Interventions: Biological: RSV vaccine GSK3003899A (formulation 6)
- Group Placebo 1 (Placebo Comparator): Subjects in this group will receive a single dose of placebo
  Interventions: Drug: Placebo comparator
- Group Placebo 2 (Placebo Comparator): Subjects in this group will receive a single dose of placebo
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Biological: RSV vaccine GSK3003892A (formulation 1) — Intramuscular (IM) vaccination in the deltoid region of the non-dominant arm at Day 0 according to protocol schedule
  Arms: Group A
Biological: RSV vaccine GSK3003893A (formulation 2) — Intramuscular (IM) vaccination in the deltoid region of the non-dominant arm at Day 0 according to protocol schedule
  Arms: Group B
Biological: RSV vaccine GSK3003895A (formulation 3) — Intramuscular (IM) vaccination in the deltoid region of the non-dominant arm at Day 0 according to protocol schedule
  Arms: Group C
Biological: RSV vaccine GSK3003896A (formulation 4) — Intramuscular (IM) vaccination in the deltoid region of the non-dominant arm at Day 0 according to protocol schedule
  Arms: Group D
Biological: RSV vaccine GSK3003898A (formulation 5) — Intramuscular (IM) vaccination in the deltoid region of the non-dominant arm at Day 0 according to protocol schedule
  Arms: Group E
Biological: RSV vaccine GSK3003899A (formulation 6) — Intramuscular (IM) vaccination in the deltoid region of the non-dominant arm at Day 0 according to protocol schedule
  Arms: Group F
Drug: Placebo comparator — Intramuscular (IM) vaccination in the deltoid region of the non-dominant arm at Day 0 according to protocol schedule
  Arms: Group Placebo 1; Group Placebo 2

SUMMARY:
The purpose of this first time in human (FTiH) study is to evaluate the safety, reactogenicity and immunogenicity of several formulations of Respiratory Syncytial Virus (RSV) investigational vaccines in healthy men.

DETAILED DESCRIPTION:
This protocol posting has been updated following protocol amendment 3 to amend the respective exclusion criterion as to only exclude subjects with clinically significant hematological/ biochemical abnormalities as per opinion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* A male between, and including, 18 and 44 years of age at the time of vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after vaccination, with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before or after vaccination.
* Previous vaccination against RSV.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the vaccine dose. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of or current autoimmune disease.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Hypersensitivity to latex.
* Any clinically significant hematological (hemoglobin level, white blood cell [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine) abnormality as per the opinion of the investigator, based on the local laboratory normal ranges.

  * Subjects with hematological/ biochemical values out of normal range which are expected to be temporary may be re-screened at a later date.
* Any acute or chronic, clinically significant disease, as determined by physical examination or laboratory screening tests.
* Malignancies within previous 5 years (excluding non-melanoma skin cancer) and lymphoproliferative disorders.
* Current alcoholism and/or drug abuse.
* Acute disease and/or fever at the time of Screening.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C /100.4°F on rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhea) without fever may be enrolled at the discretion of the investigator.
  * Subjects with acute disease and/ or fever at the time of Screening may be re screened at a later date.
* Planned move to a location that will prohibit participating in the trial until study end.
* Any other condition that the investigator judges may interfere with study procedures (e.g. drawing blood) or findings (e.g. immune response).

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2013-07-22 (Actual); Primary Completion 2014-04-09 (Actual); Study Completion 2015-03-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of each solicited local and general adverse event (AE) | During the 7 days (Days 0-6) follow-up period after vaccination
Occurrence of any hematological (hemoglobin level, white blood cells [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality | At Day 0
Occurrence of any hematological (hemoglobin level, white blood cells [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality | At Day 7
Occurrence of any hematological (hemoglobin level, white blood cells [WBC], lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality | At Day 30
Occurrence of any hematological (hemoglobin level, WBC, lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (alanine amino-transferase [ALT], aspartate amino-transferase [AST] and creatinine) laboratory abnormality | At Day 60
Occurrence of any unsolicited AE | During a 30-day (Days 0-29) follow-up period after vaccination
Occurrence of any Serious Adverse Events (SAEs) | From Day 0 to Day 60

SECONDARY OUTCOMES:
Humoral immune response in terms of neutralizing antibody titers to the investigational RSV vaccines, in all subjects, in all groups | At pre-vaccination (Day 0) and post-vaccination (Day 7, Day 30 and Day 60)
Persistence of the humoral immune response in terms of neutralizing antibody titers to the investigational RSV vaccines, in all subjects, in all groups | At Day 180 and Day 360
Occurrence of any hematological (hemoglobin level, WBC, lymphocyte, neutrophil, eosinophil and platelet count) and biochemical (ALT, AST and creatinine) laboratory abnormality | At Day 180 and Day 360
Occurrence of any SAE | From Day 60 to the study conclusion (i.e. Day 360)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Canada (3):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Toronto, Ontario

REFERENCES:
- [Derived] Steff AM, Cadieux-Dion C, de Lannoy G, Prato MK, Czeszak X, Andre B, Ingels DC, Louckx M, Dewe W, Picciolato M, Maleux K, Fissette L, Dieussaert I. Hamster neogenin, a host-cell protein contained in a respiratory syncytial virus candidate vaccine, induces antibody responses in rabbits but not in clinical trial participants. Hum Vaccin Immunother. 2020 Jun 2;16(6):1327-1337. doi: 10.1080/21645515.2019.1693749. Epub 2020 Jan 17. PMID 31951765
- See also: Results for study 116969 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/116969?search=study&b%22b''%22#rs